CLINICAL TRIAL: NCT05398315
Title: Testing the Efficacy of Interactive Alcohol Decision-Making Program
Brief Title: Interactive Alcohol Decision-Making Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Emily Grekin, Associate Professor, Wayne State University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-01-4352
Record Dates: First submitted 2022-05-19; First posted 2022-05-31 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Heavy Drinking
Keywords: Alcohol; Common Factors; Motivational Interviewing; Factorial Design

STUDY DESIGN:
Intervention Model Description: Four intervention components will be manipulated in a full factorial design, such that each participant either does or does not receive each intervention component.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be randomly assigned to a condition by a computer program. The entire study will take place online. Participants will not be aware of the condition they are in until after the study ends. Investigators/outcome assessors will only see de-identified data and will have no contact with participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Empathic Statements, MI, Male, No Backstory (Experimental): Presence of empathic statements and MI techniques. Male narrator. No narrator backstory.
  Interventions: Behavioral: Empathic Statements/Reflections; Behavioral: Male Narrator; Behavioral: MI Techniques
- No Empathic Statements, No MI, Female, No Backstory (Experimental): No empathic statements, MI techniques or narrator backstory. Female narrator
  Interventions: Behavioral: Female Narrator
- No Empathic Statements, No MI, Female, Backstory (Experimental): No empathic statements or MI techniques. Presence of narrator backstory. Female narrator
  Interventions: Behavioral: Narrator Backstory; Behavioral: Female Narrator
- Empathic Statements, MI, Female, Backstory (Experimental): Presence of empathic statements, MI techniques and narrator backstory. Female narrator
  Interventions: Behavioral: Empathic Statements/Reflections; Behavioral: Narrator Backstory; Behavioral: Female Narrator; Behavioral: MI Techniques
- No Empathic Statements, No MI, Male, No Backstory (Experimental): No empathic statements, MI techniques or narrator backstory. Male narrator
  Interventions: Behavioral: Male Narrator
- Empathic Statements, MI, Male, Backstory (Experimental): Presence of empathic statements, MI techniques and narrator backstory. Male narrator.
  Interventions: Behavioral: Empathic Statements/Reflections; Behavioral: Narrator Backstory; Behavioral: Male Narrator; Behavioral: MI Techniques
- No Empathic Statements, MI, Female, Backstory (Experimental): Presence of MI techniques and narrator backstory. No empathic statements. Female narrator.
  Interventions: Behavioral: Narrator Backstory; Behavioral: Female Narrator; Behavioral: MI Techniques
- Empathic Statements, No MI, Male, No Backstory (Experimental): Presence of empathic statements. No MI techniques or narrator backstory. Male narrator.
  Interventions: Behavioral: Empathic Statements/Reflections; Behavioral: Male Narrator
- No Empathic Statements, MI, Male, Backstory (Experimental): Presence of MI techniques and narrator backstory. No empathic statements. Male narrator.
  Interventions: Behavioral: Narrator Backstory; Behavioral: Male Narrator; Behavioral: MI Techniques
- Empathic Statements, No MI, Female, No Backstory (Experimental): Presence of empathic statements. No MI techniques or narrator backstory. Female narrator.
  Interventions: Behavioral: Empathic Statements/Reflections; Behavioral: Female Narrator
- Empathic Statements, MI, Female, No Backstory (Experimental): Presence of empathic statements and MI techniques. Female narrator. No narrator backstory.
  Interventions: Behavioral: Empathic Statements/Reflections; Behavioral: Female Narrator; Behavioral: MI Techniques
- No Empathic Statements, No MI, Male, Backstory (Experimental): Presence of narrator backstory. No empathic statements or MI techniques. Male narrator.
  Interventions: Behavioral: Narrator Backstory; Behavioral: Male Narrator
- Empathic Statements, No MI, Female, Backstory (Experimental): Presence of empathic statements and narrator backstory. No MI techniques. Female narrator.
  Interventions: Behavioral: Empathic Statements/Reflections; Behavioral: Narrator Backstory; Behavioral: Female Narrator
- Empathic Statements, No MI, Male, Backstory (Experimental): Presence of empathic statements and narrator backstory. No MI techniques. Male narrator.
  Interventions: Behavioral: Empathic Statements/Reflections; Behavioral: Narrator Backstory; Behavioral: Male Narrator
- No Empathic Statements, MI, Female, No Backstory (Experimental): Presence of MI techniques. No empathic statements or narrator backstory. Female narrator.
  Interventions: Behavioral: Female Narrator; Behavioral: MI Techniques
- No Empathic Statements, MI, Male, No Backstory (Experimental): Presence of MI techniques. No empathic statements or narrator backstory. Male narrator.
  Interventions: Behavioral: Male Narrator; Behavioral: MI Techniques

INTERVENTIONS:
Behavioral: Empathic Statements/Reflections — Presence of Empathic Statements
  Arms: Empathic Statements, MI, Female, Backstory; Empathic Statements, MI, Female, No Backstory; Empathic Statements, MI, Male, Backstory; Empathic Statements, MI, Male, No Backstory; Empathic Statements, No MI, Female, Backstory; Empathic Statements, No MI, Female, No Backstory; Empathic Statements, No MI, Male, Backstory; Empathic Statements, No MI, Male, No Backstory
Behavioral: Narrator Backstory — Presence of a narrator backstory
  Arms: Empathic Statements, MI, Female, Backstory; Empathic Statements, MI, Male, Backstory; Empathic Statements, No MI, Female, Backstory; Empathic Statements, No MI, Male, Backstory; No Empathic Statements, MI, Female, Backstory; No Empathic Statements, MI, Male, Backstory; No Empathic Statements, No MI, Female, Backstory; No Empathic Statements, No MI, Male, Backstory
Behavioral: Male Narrator — Presence of a male narrator
  Arms: Empathic Statements, MI, Male, Backstory; Empathic Statements, MI, Male, No Backstory; Empathic Statements, No MI, Male, Backstory; Empathic Statements, No MI, Male, No Backstory; No Empathic Statements, MI, Male, Backstory; No Empathic Statements, MI, Male, No Backstory; No Empathic Statements, No MI, Male, Backstory; No Empathic Statements, No MI, Male, No Backstory
Behavioral: Female Narrator — Presence of a female narrator
  Arms: Empathic Statements, MI, Female, Backstory; Empathic Statements, MI, Female, No Backstory; Empathic Statements, No MI, Female, Backstory; Empathic Statements, No MI, Female, No Backstory; No Empathic Statements, MI, Female, Backstory; No Empathic Statements, MI, Female, No Backstory; No Empathic Statements, No MI, Female, Backstory; No Empathic Statements, No MI, Female, No Backstory
Behavioral: MI Techniques — Presence of MI techniques
  Arms: Empathic Statements, MI, Female, Backstory; Empathic Statements, MI, Female, No Backstory; Empathic Statements, MI, Male, Backstory; Empathic Statements, MI, Male, No Backstory; No Empathic Statements, MI, Female, Backstory; No Empathic Statements, MI, Female, No Backstory; No Empathic Statements, MI, Male, Backstory; No Empathic Statements, MI, Male, No Backstory

SUMMARY:
This project aims to develop a maximally effective, computer-delivered brief intervention (CDBI) for reducing heavy alcohol use. More specifically, the investigators will examine outcomes of different versions of a CDBI in which the presence/absence of empathic statements, the gender of the narrator, the presence/absence of a narrator backstory, and the use/non-use of motivational interviewing techniques are systematically manipulated using a factorial design. Participants (352 heavy drinkers) will be randomly assigned to 1 of 16 intervention conditions, representing all combinations of the 4 variables being manipulated. The investigators hypothesize that there will be significant main effects of all four factors being manipulated on (a) subjective reactions to the CDBI and (b) alcohol outcomes at 1-month follow-up

DETAILED DESCRIPTION:
The National Survey on Drug Use and Health estimates that 19.3 million individuals ages 12 and over met criteria for an alcohol use disorder in the past year, fully 87.4% of whom neither received any treatment in the past 12 months, nor wanted it. Recognition of this tremendous gap has led to efforts, both nationally and internationally, to implement proactive screening and brief intervention. Brief interventions have proven efficacious in reducing unhealthy drinking with effect sizes in meta-analyses ranging from small to moderate. Brief interventions are also uniquely applicable to non-treatment-seeking populations, who may refuse extended treatment but accept a minimal, opportunistic intervention. However, the public health impact of brief interventions has been limited by substantial difficulty with implementation. Further, positive overall findings in meta-analyses obscure the results of multiple rigorous efficacy trials showing no brief intervention effect on alcohol use. Both of these issues-the implementation challenges and the inconsistency in outcomes-suggest that changes are needed before brief alcohol interventions can meet their full potential.

Technology offers exciting potential in both respects. First, computer-delivered brief interventions (CDBIs) can be presented inexpensively, with perfect fidelity, and without the need for training or provider time. Second, their replicability, flexibility, and modularity makes them the perfect platform for (a) isolating the active ingredients that are associated with positive outcomes; and thereby (b) continually optimizing CDBIs to achieve cumulative increases in efficacy.

The overall goal of this research is to develop a maximally effective and replicable CDBI for reducing heavy alcohol use. To accomplish this, the investigators will use the Multiphase Optimization Strategy (MOST), an efficient method for optimizing intervention content that uses factorial designs to evaluate main and interaction effects of specific intervention components. The selection of components will be guided by: (a) Common Factors Theory, which highlights the tremendous contribution of relational factors, such as empathy, alliance and positive regard to therapy outcomes, but which is of unknown relevance to CDBIs; and (b) the Media Equation Theory, which suggests that people automatically respond to computers in social ways, particularly when those computers replicate human characteristics. Guided by this literature, the investigators will examine outcomes of a CDBI in which empathic statements, the gender of the narrator, the presence/absence of a narrator backstory, and the use/non-use of motivational interviewing techniques are systematically manipulated using a factorial design.

Specific aims are as follows:

1. Develop 16 distinct, time-consistent, computer-delivered sessions representing all possible combinations of the following four factors (each of which will be binary; i.e. either present vs. absent or male vs. female): (1) narrator gender, (2) empathic statements and reflections, (3) narrator backstory, and (4) use of motivational techniques.
2. Evaluate main and interaction effects of the five factors by randomly assigning 352 heavy drinkers to the 16 sessions (each of the four factors being presented to half of the participants) and evaluating (1) subjective reactions to the CDBI at baseline and (2) alcohol use at 1-month follow-up.

Hypothesis 1. Subjective reactions to the CDBI, disclosure of alcohol use and consequences, and motivation to reduce alcohol use will be higher and alcohol use at follow-up will be lower in the presence of (1) empathic statements, (2) a narrator backstory and (3) motivational techniques. The effects of narrator gender will be examined in an exploratory way (i.e., no a priori hypotheses).

Hypothesis 2. Subjective reactions will be more positive, disclosure and motivation to reduce alcohol use will be higher, and alcohol use at follow-up will be lower when the two relational factors (empathy and narrator backstory) are combined with the presence of motivational content.

ELIGIBILITY:
Inclusion Criteria:

* Over age 18
* Access to the internet.
* Males must consume at least 14 drinks per week or 4 drinks per day
* Females must consume at least 7 drinks per week or 3 drinks per day

Exclusion Criteria:

* Under age 18
* No internet access
* Males who consume less than 14 drinks per week or 4 drinks per day
* Females who consume less than 7 drinks per week or 3 drinks per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Quantity and Frequency of Alcohol Use | Given pre-intervention and at 1-month follow-up
  The Timeline Followback Questionnaire (TLFB) will be given to assess past month alcohol use.
Change in Alcohol-Related Consequences | Given pre-intervention and at 1-month follow-up
  Assessed with the Brief Young Adult Alcohol Consequences Questionnaire which assess the occurrence/ non-occurrence of 24 alcohol consequences.
Participant Satisfaction with the Intervention | Given immediately after completing the intervention
  Fifteen item measure assessing how much participants liked the intervention and felt respected by it.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Grekin, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grekin ER, Thomas HA, Ondersma SJ. Testing the efficacy of narrator empathy, self-disclosure, gender, and use of brief motivational interviewing techniques in a brief internet-based intervention for alcohol use. Psychol Addict Behav. 2024 May;38(3):231-242. doi: 10.1037/adb0001003. Epub 2024 Mar 14. PMID 38483522